CLINICAL TRIAL: NCT02975492
Title: Evaluation de l'Impact d'un Mode de supplémentation en Vitamine D (Dose séquentielle vs Dose Quotidienne) Sur l'Incidence de l'Hypercalciurie Chez Des Sujets Des départements du Gard et de l'Hérault agés de 2 à 18 Ans. Etude contrôlée randomisée en 2 Groupes parallèles
Brief Title: Assessing the Impact of a Mode of Vitamin D Supplementation (Sequential Dose vs Daily Dose) on the Incidence of Hypercalciuria in Subjets Aged From 2 to 18 Years
Acronym: DonneDVit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL15_0500; UF 9676 (Other: Montpellier University Hospital)
Record Dates: First submitted 2016-11-07; First posted 2016-11-29 (Estimated); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Transient Hypercalciuria
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cholecalciferol sequential dose (Experimental): cholecalciferol : 100 000 Unit International (UI), sequential dose (2 mL)
  Interventions: Drug: Cholecalciferol sequential dose
- Cholecalciferol daily dose (Experimental): cholecalciferol : 1000 UI, daily dose during 28 days (0.1 ml by day)
  Interventions: Drug: Cholecalciferol daily dose

INTERVENTIONS:
Drug: Cholecalciferol sequential dose — sequential dose administration of the treatment
  Other Names: Vitamin D
  Arms: Cholecalciferol sequential dose
Drug: Cholecalciferol daily dose — daily dose administration of the treatment
  Other Names: Vitamin D
  Arms: Cholecalciferol daily dose

SUMMARY:
Recommendations for vitamin D supplementation for subjets between 2 and 18 years offer strong sequential doses of vitamin D: 2 times 100 000 units in spaced winter period of 3 months. Data from the literature show a further increase in the incidence of oxalo-calcium stones in children and adolescents associated with hypercalciuria with training Randall plates, essential step lithogenesis calcium oxalate. Knowing the links between vitamin D and urinary calcium excretion, these data lead to the question of increased sensitivity in some children with vitamin D, sensitivity could explain these situations with hypercalciuria increase the gallstone risk. This increased sensitivity to vitamin D may unmask particularly if inputs of high doses of vitamin responsible then a transient hypercalciuria with development of microcrystals.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 to 17 years included
* Obtaining informed consent of the parents signed
* Participants aged 18 years included

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 280 (Estimated)
Dates: Start 2017-12-14 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes from calcium level in urines at day 7, day 14 and day 28 | day 7, day 14 and day 28

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Pediatric department, Montpellier
  - Pediatric department, Nîmes

IPD SHARING:
Plan to Share IPD: No